CLINICAL TRIAL: NCT03892083
Title: Effect of Transcranial Direct Current Stimulation (tDCS) on Postural Control of Children With Developmental Coordination Disorder: a Double-blind Randomized Controlled Trial
Brief Title: Effect of tDCS on Postural Control of Children With DCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 39398214.4.3001.5391
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-03

CONDITIONS: Developmental Coordination Disorder
Keywords: Developmental coordination disorder; Postural balance; Transcranial Direct Current Stimulation; Children; Child Development
MeSH Terms: conditions — Motor Skills Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Anodal tDCS (M1) (Active Comparator): tDCS applied over primary motor cortex. Dose: 1mA, 20 minutes
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Anodal Cerebellar tDCS (Experimental): tDCS applied over the cerebellum. Dose: 1mA, 20 minutes
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Cathodal Cerebellar tDCS (Experimental): tDCS applied over the cerebellum. Dose: 1mA, 20 minutes
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Sham tDCS (Sham Comparator): tDCS applied over the cerebellum Dose: 1mA, 20 minutes (30s ON)
  Interventions: Device: Transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — Transcranial direct current stimulation is a noninvasive technique of neuronal modulation that has been used in different neurological conditions, including children with cerebral palsy.

SUMMARY:
This study investigates the effects of Transcranial Direct Current Stimulation (tDCS) on postural control of children with Developmental Coordination Disorder (DCD). All participants will receive four conditions of stimulation, in a crossover protocol: cerebellar anodic, cerebellar cathodic, primary motor cortex anodic (M1) or sham tDCS.

DETAILED DESCRIPTION:
Developmental Coordination Disorder (DCD) is a highly frequent neurodevelopmental disorder with negative impacts on children's motor repertoire, quality of life and general health. One of the main problems faced is the balance deficit, which although well characterized in this population, little is known about the etiological core of this impairment. The cerebellum appears to be a functionally impaired structure in DCD, but frontal motor areas are also involved. Transcranial Direct Current Stimulation (tDCS) is a noninvasive way of inducing local-specific polarity-dependent synaptic modulation. Cerebellar tDCS (CE-tDCS) is even more recent, with still unclear results on its effects on postural balance, with only one study in children, which requires us to better understand the type of stimulation necessary to induce balance improvement in children with DCD.

Thus, the investigators aimed to verify the effects of anodal tDCS over primary motor cortex (M1-atDCS) and CE-tDCS (anodic, cathodic and sham) on the balance of children with DCD, compared to children without DCD.

METHODS: Fifteen children with DCD (total MABC-2 and balance <15%, with DCDQ positive / TL positive) and 15 children without DCD (MABC-2 total and balance ≥50% and DCDQ negative) will be assessed by platform stabilometry (PS) before and after receiving M1, cerebellar anodic, cerebellar cathodic, primary motor cortex anodic (M1) or sham tDCS (crossover). They will be evaluated under conditions without proprioceptive manipulation (direct on PS) with open and closed eyes, and with proprioceptive manipulation (on foam surface) with open and closed eyes.

ELIGIBILITY:
Inclusion Criteria:

* children of both sex, aged between seven years 0 months and 10 years and 11 months;
* Assent of the child by the Term of Assent and acceptance of parents and / or guardians to participate in the study by signing the Free and Informed Consent Form;
* Children with DCD indicative according to DSM-5 presenting Percentile <15 in the MABC-2 Motor Evaluation Battery and in the balance domain; and the score indicated for each age by the Developmental Coordination Disorder Questionnaire DCDQ-Brazil (TDC Group).
* Children without DCD presenting Percentile ≥ 50 in the total score and in the MABC-2 Motor Assessment Battery Balance domain, without indicative by DCDQ (Control Group - GC).
* Absence of intellectual disability considering performance above the 25th percentile on the RAVEN Color Progressive Matrix scale
* Absence of visual or auditory deficiencies; cardiopathies; rheumatic or orthopedic dysfunctions; neurological or psychiatric problems (except ADHD and language disorder because they are the most comorbid disorders with DCD).

Exclusion Criteria:

• Signs of excessive discomfort during or after any procedures or sessions involved in the research.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Change from COP - AP axis | Baseline and Post-tDCS (immediately after tDCS)
  Postural instability will be evaluated using a force plate to record center of pressure displacement (COP) in antero-posterior (AP) axis in centimeters
Change from COP - ML axis | Baseline and Post-tDCS (immediately after tDCS)
  Postural instability will be evaluated using a force plate to record center of pressure displacement (COP) in Mediolateral (ML) axis in centimeters
Change from COP - area | Baseline and Post-tDCS (immediately after tDCS)
  Postural instability will be evaluated using a force plate to record center of pressure displacement (COP) area (cm²)

OTHER OUTCOMES:
Adverse effects | Immediately after tDCS
  Adverse effects will be evaluated using structured questionnaire.
  Active collection uses a questionnaire with records of the duration (minutes or hours) and intensity (Numerical Rating Scale 0-10) of adverse symptoms reported by the patient.
  Complaints:
  Headache Scalp pain Tingling Itching Redness Burning sensations Sleepiness Trouble concentrating Nausea Mood change

CONTACTS AND LOCATIONS:
Overall Officials: Renata H Hasue, pHD, Principal Investigator — Faculty of Medicine, University of São Paulo
Locations (1):
- Department of Physical Therapy, Communication Sciences and Disorders, and Occupational Therapy, Faculty of Medicine, University of São Paulo, São Paulo, Brazil